CLINICAL TRIAL: NCT03081065
Title: Nutritional Intervention With Mediterranean Diet in the Prevention of Recurrence of Depression
Brief Title: Mediterranean Diet and Recurrence of Depression
Acronym: PREDI-DEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Las Palmas de Gran Canaria (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Almudena Sanchez-Villegas, Professor of Preventive Medicine, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ULPGC
Record Dates: First submitted 2017-02-06; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Clinical Trial; Depression; Mediterranean, Diet
MeSH Terms: conditions — Depression | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet+ extra virgin olive oil (Experimental): Free supply with extra virgin olive oil and nuts plus educational advice
  Interventions: Dietary Supplement: Mediterranean Diet
- Mediterranean Diet+ tree nuts (Experimental): Free supply with tree nuts plus educational advice
  Interventions: Dietary Supplement: Mediterranean Diet
- Control (No Intervention): Usual care

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — Nutritional advice to follow a Mediterranean diet and supplementation with extra virgin olive oil and nuts
  Arms: Mediterranean Diet+ extra virgin olive oil; Mediterranean Diet+ tree nuts

SUMMARY:
OBJECTIVES:To assess the effect of the intervention with Mediterranean Diet (MD) supplemented with extra virgin olive oil (EVOO) or tree nuts (TN) during 2 years (compared to a control group without intervention) on the risk of recurrence of unipolar depressive disorder in patients with partial or total remission for unipolar depressive disorder (1). Differences between groups in changes in residual symptoms (2), quality of life (QL) (3), biochemical parameters (4) and in the risk of medical/psychiatric co-morbidities (5) will be also analyzed. Finally, gut microbiota and its changes will be collected and compared between groups (6). METHODS: Multicenter clinical trial with 3 arms of intervention (MD+EVOO; MD+TN;control) during 2 years. Adults with previous episodes of unipolar depressive disorder in partial or total remission stage (determined through Montgomery-Asberg questionnaire and MINI interview) will be included. Participants with current depression, psychiatric co-morbid disorders or with problems to follow dietary recommendations will be excluded. A recurrence ratio of 35% in the MD groups and of 50% in the control group will be considered (Hazard Ratio: 0.7). We estimate a sample size of 720 participants (750 to count for losses) (90% power and 5% alpha error). Intervention will be performed through postal mail (recipes and information), email, phone y new technologies (Web page/mobile app) with periodic contacts with psychiatrics and dieticians and postal mail for free EVOO and nuts supply. Information from participants will be gathered with validated questionnaires of diet, physical activity, QL, or symptoms using postal mail, email, Web page or the phone. The analyses will be performed by intention to treat.

DETAILED DESCRIPTION:
DESIGN This trial is a multicenter, parallel clinical trial with 3 intervention arms, two of them with Mediterranean Diet (MD) supplemented extra virgin olive oil (EVOO) or tree nuts (TN) and the last one is the control group without any kind of nutritional intervention.

SAMPLE Seven groups across Spain have agreed to participate in the trial and will recruit participants. With a 5% alpha error, 90% power and considering an incidence of recurrence of depression after 2 years of intervention of 35% in the MD groups and of 50% in the control group, we will need 240 participants in each group. Considering also possible losses, finally we have estimated a sample size of 750 participants, 108 participants in each of the recruitment centers.

The inclusion criteria were defined after an exhaustive review of the scientific literature and under consensus among all the psychiatric and clinical psychologists included in the study. We will include 1 participant with a unique episode of depression for each three participants with 2 or more episodes.

SELECTION OF PARTICIPANTS Clinical psychologists and psychiatrists will carry out the pre-selection of the participants after a detailed review of their clinical records. When a participant is pre-selected, the psychiatrists will perform a semi-structured interview (MINI interview) according to DSM-V criteria and a Montgomery-Asberg Depression Rating Scale to discard depression and other mental disorders diagnoses and to assess depression remission degree. This information will be completed with some questions included in the eligibility questionnaire such as medical conditions or problems related with the adherence to the MD. Moreover, participants will receive detailed written information of the study and the informed consent that they have to sign. The nurse will perform a venipuncture to obtain a blood sample according to the normal protocol. Moreover, in a subsample of the sample the participants will be instructed to collect a stool sample. Finally, all the data will be transferred to the dietitians of the study.

The dietitians of the study will be responsible for the periodic contact with the participants and to perform the nutritional intervention and follow-up. Contacts will be made through new technologies such as a web platform, a mobile app, telephone and email. Additionally, if a participant is not familiarized with these technologies, the dieticians will use postal mail to send all the information.

RANDOMIZATION AND INTERVENTION The study dietitians will perform the randomization of the participants to the corresponding intervention group following tables of random allocation according to the recruitment order balanced by age, group, and recruitment center. The randomization process will be performed from the coordination center. The psychiatrists who will perform mental evaluation of the participants will not participate in the process of randomization to avoid knowing to which group has been assigned each patient.

MD groups The protocol used in this trial is similar to that applied in the PREDIMED trial. In fact, the dietitians of this trial have participated in the PREDIMED trial and are collaborating also in the PREDIMED-PLUS.

The MD group will receive EVOO (A 1-liter free supply every 2 weeks) or TN (20 grams per day).

In the beginning of the trial the dietitian will provide a comprehensive number of reasons to adopt a MD to each participant, and will negotiate a change in his/her diet, working with the subject to determine what he or she considers an attainable goal. This compliance degree will be assessed every 3 months by the dietician through a telephone call to the participants. Every 3 months participants will also receive information about food items typical of the MD and adapted to the season of the year, a quantitative 1-week buying list of food items according to the season of the year, a weekly plan of meals (with detailed menus) adapted to the buying list and cooking recipes for cuisine practices according to the suggested menus.

Web page and mobile app will be updated each week with news related MD and its health effects.

Any doubt or suggestion made by our participants will be taken into account by our dietitians at any moment of the intervention period.

Control group Control group will not receive any kind of nutritional intervention although these participants will have an email and access to the project web page but with some limits for contents related with the intervention. To avoid losses during follow-up in the group, these participants will receive some incentives such as cinema tickets or discount vouchers in supermarkets

INFORMATION ASSESSMENT

1. MINI interview To assess mental disorders diagnosis
2. Montgomery-Asberg Depression Rating Scale questionnaire (Med Clin 2002;118:493-9) To assess depressive symptoms severity
3. Eligibility questionnaire: to assess presence of severe diseases, food allergies and assessment of the willingness to make diet changes (Prochaska model)
4. Baseline general and follow-up questionnaires: Socio-economic, anthropometric and life-style variables and diagnosis of diseases and use of psychotherapy and medication
5. Conformity to the Mediterranean diet questionnaire (J Nutr 2011; 141:1140-5)
6. Semi-quantitative food frequency questionnaire (Br J Nutr 2010;103:1808-16)
7. Minnesota physical activity questionnaire (Am J Epidemiol 1994;139:1197-209)
8. SF-36 quality of life questionnaire (Gac Sanit 2005;19 :135-50)

A clinical interview will be administered to discard a diagnosis of depression at baseline. This interview will be repeated every year. Coinciding with the medical visit blood extraction will be performed every year. Stool samples will be collected in a subsample both in the beginning and at the end of the trial.

Every four months psychiatrists will administer the Montgomery-Asberg questionnaire by telephone except in the beginning of the study or once a year in which the questionnaire will administer face to face in the consulting room. If there is any suspicion of depression reported by the psychiatrist after the telephone interview or reported by any patient relative the participants will be cited to attend the consulting room.

The adherence to the MD, nutrient and food intake, physical activity and quality of life will be assessed through validated questionnaires that were already used in the PREDIMED trial. The dietitians will collect information on diet, physical activity, quality of life and medical and life-style variables at baseline and yearly using new technologies, and the telephone.

ELIGIBILITY:
Inclusion Criteria:

* adults
* with a previous diagnosis of depression in the last 5 years and in a stage of total or partial remission

Exclusion Criteria:

* presence of comorbid psychiatric disorders (anxiety, bipolar disorder, personality disorders, alcohol and drug abuse, mania, psychosis)
* presence of severe medical condition with survival lower than one year)
* history of food allergy with hypersensitivity to any of the components of olive oil or nuts
* presence of disorders of chewing or swallowing
* difficulties to change dietary habits
* institutionalized patients and those participants who lack autonomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2017-03-20 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Time until recurrence of depression (defined as a clinical diagnosis of unipolar depressive disorder made by a Psychiatrist from the research team) | From date of randomization until the date of first documented depressive episode diagnosis assessed up to 32 months
  New diagnoses of episodes of depression (recurrent depression as participants have a history of unipolar depressive disorder).

SECONDARY OUTCOMES:
Change in depressive symptoms using the Montgomery Asberg Depression Rating Scale | Yearly (baseline, 1-year, 2-year of follow-up)
  Short (from baseline to the 1st-y) and long (from baseline to the 2nd-y) changes in depressiove symptoms (quantitative measure)
Change in quality of life using the SF-36 quality of life questionnaire | Yearly (baseline, 1-year, 2-year of follow-up)
  Short (from baseline to the 1st-y) and long (from baseline to the 2nd-y) changes in the eight domains (4 physical and 4 mental domains) of the SF-36 questionnaire
Change in biochemical parameters (plasma levels of total cholesterol, HDL-cholesterol, LDL-cholesterol, glucose, protein C Reactive) | Yearly (baseline, 1-year, 2-year of follow-up)
  Short (from baseline to the 1st-y) and long (from baseline to the 2nd-y) changes in biochemical parameters
Change in microbiota in stool samples | Change from baseline to the second year of follow-up
  Gut microbial diversity and DNA analysis and their changes during the trial
Incidence of physical diseases (Clinically confirmed after an exhaustive review of clinical records of the participants) | From date of randomization until the date of first documented physical disease diagnosis assessed up to 32 months
  New diagnoses of medical diseases (mainly cancer, cardiovascular disease, metabolic syndrome or diabetes) reported by the participants in the follow-up questionnaires (later confirmed)
Incidence of other psychiatric disorders (clinical diagnosis made by a Psychiatrist from the research team) | From date of randomization until the date of first documented psychiatric disorder diagnosis assessed up to 32 months
  New diagnoses of psychiatric disorders made by a psychiatrist during the follow up period (bipolar disorder, schizophrenia, personality disorder, mania, eating disorders, drug abuse and anxiety disorder)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabrera-Suarez BM, Lahortiga-Ramos F, Sayon-Orea C, Hernandez-Fleta JL, Gonzalez-Pinto A, Molero P, Vega-Perez R, Sanchez-Villegas A; PREDI-DEP investigators. Effect of a dietary intervention based on the Mediterranean diet on the quality of life of patients recovered from depression: Analysis of the PREDIDEP randomized trial. Exp Gerontol. 2023 May;175:112149. doi: 10.1016/j.exger.2023.112149. Epub 2023 Mar 20. PMID 36933773
- [Derived] Cabrera-Suarez B, Pla J, Gonzalez-Pinto A, Hernandez J, Chiclana-Actis C, Ortuno F, Florido-Rodriguez M, Sanchez-Villegas A, Investigators PD. 'Effectiveness of a remote nutritional intervention to increase the adherence to the Mediterranean diet among recovered depression patients'. Nutr Neurosci. 2023 Aug;26(8):696-705. doi: 10.1080/1028415X.2022.2081448. Epub 2022 Jul 11. PMID 35816397
- [Derived] Sanchez-Villegas A, Cabrera-Suarez B, Molero P, Gonzalez-Pinto A, Chiclana-Actis C, Cabrera C, Lahortiga-Ramos F, Florido-Rodriguez M, Vega-Perez P, Vega-Perez R, Pla J, Calvino-Cabada MJ, Ortuno F, Navarro S, Almeida Y, Hernandez-Fleta JL. Preventing the recurrence of depression with a Mediterranean diet supplemented with extra-virgin olive oil. The PREDI-DEP trial: study protocol. BMC Psychiatry. 2019 Feb 11;19(1):63. doi: 10.1186/s12888-019-2036-4. PMID 30744589